CLINICAL TRIAL: NCT01777997
Title: A Prospective, Single-Arm, Open-Label Study to Evaluate the Effect of Fixed-Dose Emtricitabine/Rilpivirine/Tenofovir Disoproxil Fumarate on T-Cell Activation, Absolute CD4+ T-Cell Count, Inflammatory Biomarkers and Viral Reservoir in Treatment-Naïve HIV-1 Controllers
Brief Title: FTC/RPV/TDF on T-Cell Activation, CD4+ T-Cell Count, Inflammatory Biomarkers and Viral Reservoir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5308; 1U01AI068636 (NIH)
Record Dates: First submitted 2013-01-10; First posted 2013-01-29 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2017-12

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Emtricitabine; Emtricitabine, Rilpivirine, Tenofovir Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FTC/RPV/TDF (Experimental)
  Interventions: Drug: Emtricitabine/rilpivirine/tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Emtricitabine/rilpivirine/tenofovir disoproxil fumarate — Step 1: From entry through week 12, the participants received no study treatment. From week 12 through week 60, the participants received one fixed dose combination emtricitabine/rilpivirine/tenofovir disoproxil fumarate (FTC/RPV/TDF) tablet daily.
  Step 2 (Optional): From week 60 through week 108, the participants either received one FTC/RPV/TDF tablet daily or no study treatment.
  Other Names: FTC/RPV/TDF; Complera

SUMMARY:
This study was done with people who were infected with HIV, but did not show any signs of having HIV. They were also feeling well without taking HIV medication and had low or undetectable levels of the virus in the blood. The purpose of this study was to see if taking HIV medication (antiretroviral therapy [ART]) would reduce immune activation (a signal that the body is fighting an infection) in people who have HIV, but did not show symptoms. Also this study helped determine how safe the drug was and how well people reacted to the drug.

For this study, the following antiretroviral therapy (ART) was be provided in the form of a single tablet that contains three different drugs: emtricitabine/rilpivirine/tenofovir disoproxil fumarate (FTC/RPV/TDF). These drugs were combined as one tablet which was approved by the Food and Drug Administration (FDA) as a single pill to treat HIV infection. The HIV medication provided was one of the recommended treatments for HIV, including people with low viral loads (how much HIV you have in your body) who were taking HIV drugs for the first time. The risks seen with this HIV medication were the same that one would encounter when taking these drugs outside of the study.

DETAILED DESCRIPTION:
AIDS Clinical Trials Group (ACTG) A5308 was a single-arm clinical trial to evaluate the effect of initiating fixed-dose combination (FDC) FTC/RPV/TDF on CD8+ T-cell activation and other immunologic and virologic biomarkers among treatment-naïve HIV-1 controllers with any absolute CD4+ T-cell count. At study entry, these participants were followed off ART for a 12-week lead-in period, and then at week 12, participants initiated FDC FTC/RPV/TDF and had 48 weeks of follow-up to evaluate the primary endpoint.

All participants who completed Step 1 (48 weeks of ART) had the option to register to Step 2, for an additional 48 weeks of follow-up, and had the choice of either continuing FDC FTC/RPV/TDF or follow-up with no study treatment.

Participants underwent safety and tolerability evaluations throughout the study, including physical examinations and clinical assessments. Pregnancy tests were performed on women of childbearing potential. Collection of stored blood plasma/peripheral blood mononuclear cell (PBMC) samples occurred at entry and weeks 0, 4, 12, 24, 36, 48, 60, 72 and 96 on ART.

Only participants who were on intervention (ART) for at least 24 weeks had samples sent for testing of immunologic and virologic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

Step 1

* HIV-1 infection
* ART-naïve defined as ≤7 days of antiretroviral (ARV) treatment at any time prior to entry
* Documentation of HIV-1 RNA <500 copies/mL verified by at least two measurements prior to the screening RNA specimen
* Screening HIV-1 RNA <500 copies/mL using an US FDA-approved assay obtained within 60 days prior to study entry by any laboratory that has a CLIA certification or its equivalent
* Laboratory values obtained within 60 days prior to entry by any laboratory that has a CLIA certification or its equivalent:

  * Absolute neutrophil count (ANC) >=500/mm^3
  * Hemoglobin >=8.0 g/dL
  * Platelet count >=40,000/mm^3
  * Aspartate aminotransferase (AST) (SGOT), alanine aminotransferase (ALT) (SGPT), and alkaline phosphatase <=5 X Upper Limit of Normal (ULN)
  * Total bilirubin <=2.5 X ULN
  * Calculated creatinine clearance (CrCl) >=60 mL/min
* For females of reproductive potential, negative serum or urine pregnancy test within 48 hours prior to study entry by any clinic or laboratory that has a CLIA certification or its equivalent
* Female subjects of reproductive potential, who are participating in sexual activity that could lead to pregnancy, must agree to use at least one reliable form of contraceptive (ie, condoms (male or female) with or without a spermicidal agent; a diaphragm or cervical cap with spermicide; an intrauterine device (IUD); or hormone-based contraceptive) while receiving the protocol-specified treatment and for 6 weeks after stopping the medications
* No evidence of any exclusionary resistance mutations based on results from any genotype assay from any laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent

Step 2

* Completion of Step 1
* Ability and willingness of subject to choose to receive either open-label ART FDC (FTC/RPV/TDF) or no study treatment for an additional 48 weeks
* For females of reproductive potential, negative serum or urine pregnancy test within 48 hours prior to the week 60 visit by any clinic or laboratory that has a CLIA certification or its equivalent

Exclusion Criteria:

Step 1

* Chronic hepatitis B virus (HBV) infection (documented by hepatitis B surface antigen (HBsAg) seropositivity)
* Breastfeeding
* Use of immunomodulators (eg, interleukins, interferons, cyclosporine), topical imiquimod, HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry or plans to start immunomodulators, topical imiquimod, HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy during the study
* Known allergy/sensitivity or any hypersensitivity to components of study drug(s) or their formulation
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Acute or serious illness requiring systemic treatment and/or hospitalization within 30 days prior to entry
* Symptomatic HIV disease and/or AIDS-defining illness.
* Vaccinations within 7 days prior to study entry
* Plans to initiate hepatitis C treatment during the study
* Perinatally-acquired HIV
* Use of any of the following medications within 7 days prior to study entry:

  * St. John's wort (Hypercium perforatum)
  * Anticonvulsants (eg, oxacarbazepine, phenobarbital, phenytoin)
  * Anti-infectives (eg, rifabutin, rifampin, rifapentine)
  * Corticosteroids (eg, dexamethasone (more than 1 dose))
  * Proton pump inhibitors (eg, esomeprazole, lansoprazole, omeprazole, pantoprazole, rabeprazole)

Step 2

* Plans to start immunomodulators, topical imiquimod, HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy during Step 2 of the study
* Plans to initiate hepatitis C treatment during Step 2 of the study

NOTE: Please refer to the protocol for detailed eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-04-25 (Actual); Primary Completion 2016-02-19 (Actual); Study Completion 2017-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Li, M.D., M.M.S., Study Chair — Brigham and Women's Hospital Therapeutics (BWHT) CRS
Locations (19):
- United States (19):
  - 31788 Alabama CRS, Birmingham, Alabama
  - 801 University of California, San Francisco HIV/AIDS CRS, San Francisco, California
  - Whitman Walker Health CRS (31791), Washington D.C., District of Columbia
  - The Ponce de Leon Ctr. CRS (5802), Atlanta, Georgia
  - Northwestern University CRS (2701), Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS (2702), Chicago, Illinois
  - IHV Baltimore Treatment CRS (4651), Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS (101), Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS (107), Boston, Massachusetts
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS (31787), Rochester, New York
  - Bronx-Lebanon Hosp. Ctr. CRS (31469), The Bronx, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Moses H. Cone Memorial Hospital CRS (3203), Greensboro, North Carolina
  - University of Cincinnati CRS (2401), Cincinnati, Ohio
  - Metro Health CRS (2503), Cleveland, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS (6201), Philadelphia, Pennsylvania
  - Pitt CRS (1001), Pittsburgh, Pennsylvania
  - The Miriam Hosp. ACTG CRS (2951), Providence, Rhode Island
  - Houston AIDS Research Team CRS (31473), Houston, Texas

REFERENCES:
- See also: Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009) — http://rsc.tech-res.com/safetyandpharmacovigilance/
- See also: Requirements, definitions, and methods for expedited reporting of Adverse Events (AEs) in Version 2.0 of the DAIDS EAE Manual — http://rsc.tech-res.com/safetyandpharmacovigilance/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited at 19 Clinical Research Sites (CRSs) in the United States between April 25, 2013 and December 22, 2014.
Groups:
- FTC/RPV/TDF: Step 1: From entry through week 12, the participants received no study treatment. From week 12 through week 60, the participants received one fixed dose combination emtricitabine/rilpivirine/tenofovir disoproxil fumarate (FTC/RPV/TDF) tablet daily. Participants in the primary outcome analysis were on ART for at least 24 weeks and up to 48 weeks.
  Step 2 (Optional): From week 60 through week 108, the participants either received one FTC/RPV/TDF tablet daily or no study treatment. Participants in exploratory analyses were on ART for at least 72 weeks and up to 96 weeks.
Period: 12 Week lead-in of no ART
Arm/Group | FTC/RPV/TDF
Started | 38
Completed | 36
Not Completed | 2
Not completed — Severe debilitation | 2
Period: Weeks 0 to 24/48 on ART
Arm/Group | FTC/RPV/TDF
Started | 36
Completed | 35 (7 of these participants opted not to continue ART into next period)
Not Completed | 1
Not completed — Participant felt treatment not working | 1
Period: Weeks 48 to 72/96 on ART
Arm/Group | FTC/RPV/TDF
Started | 28
Completed | 26
Not Completed | 2
Not completed — Death | 1
Not completed — Took prohibited/precautionary meds | 1

BASELINE CHARACTERISTICS:
Population: Participants who were on intervention (ART) for at least 24 weeks
Groups:
- FTC/RPV/TDF: Step 1: From entry through week 12, the participants received no study treatment. From week 12 through week 60, the participants received one fixed dose combination emtricitabine/rilpivirine/tenofovir disoproxil fumarate (FTC/RPV/TDF) tablet daily.
  Step 2 (Optional): From week 60 through week 108, the participants either received one FTC/RPV/TDF tablet daily or no study treatment.
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 35
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [32 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 20
Race/Ethnicity, Customized [Number; unit: participants]
  White non-Hispanic | 6
  Black non-Hispanic | 26
  Hispanic (regardless of race) | 3
Region of Enrollment [Number; unit: participants]
  United States | 35
CD4+ T-cell count [Median (Inter-Quartile Range); unit: cells/mm^3] — Baseline CD4+ T-cell count is the mean of the two measurements obtained prior to the start of ART (study entry and study week 12).
  cells/mm^3 | 682 [564 to 1003]
HIV-1 RNA by Abbott Assay [Count of Participants; unit: Participants]
  Pre-ART (study entry): <40 copies/mL | 16
  Pre-ART (study entry): >=40 copies/mL | 19
  Week 0 on ART (study week 12): <40 copies/mL | 13
  Week 0 on ART (study week 12): >=40 copies/mL | 22
Percentage of CD8+ T-cells that are CD38+HLA-DR+ [Median (Inter-Quartile Range); unit: % of CD8+ T-cells] — Baseline CD8+ T-cell activation is the mean of the two measurements obtained prior to the start of ART (study entry and study week 12).
  % of CD8+ T-cells | 24.6 [19.6 to 33.4]
Percentage of CD4+ T-cells that are CD38+HLA-DR+ [Median (Inter-Quartile Range); unit: % of CD4+ T-cells] — Baseline CD4+ T-cell activation is the mean of the two measurements obtained prior to the start of ART (study entry and study week 12).
  % of CD4+ T-cells | 2.6 [2.2 to 4.1]
Interleukin (IL)-6 [Median (Inter-Quartile Range); unit: log10(pg/mL)] — Baseline IL-6 is the mean of the two log10-transformed measurements obtained prior to the start of ART (study entry and study week 12).
  log10(pg/mL) | 0.17 [0.08 to 0.38]
D-dimer [Median (Inter-Quartile Range); unit: log10(ng/mL)] — Baseline D-dimer is the mean of the two log10-transformed measurements obtained prior to the start of ART (study entry and study week 12).
  log10(ng/mL) | 2.58 [2.39 to 2.82]
Quality of life (QoL) index [Median (Inter-Quartile Range); unit: units on a scale] — QoL index was obtained by averaging the five responses on the Euro-Quality of Life questionnaire (EQ-5D), where a response of 0 indicates "no problems/no discomfort", 1 indicates "some problems/moderate discomfort" and 2 indicates "unable to perform activities/extreme discomfort". Baseline QoL index is the mean of the two averages obtained prior to the start of ART (study entry and study week 12).
  units on a scale | 0.2 [0.1 to 0.3]

OUTCOME MEASURES:

1. Primary Outcome: Change in Levels of CD8+ T-cell Activation (Defined as the Percentage HLA-DR+/CD38+) From Baseline to Weeks 24 and 48 on ART
Description: Mean change from baseline (pre-ART [study entry] and week 0 on ART [study week 12]), estimated with a repeated measures analysis (jointly to weeks 24 and 48 on ART) using generalized estimating equations (GEE)
Time Frame: From baseline (pre-ART and week 0 on ART) to weeks 24 and 48 on ART
Population: As-treated: Only participants with results while receiving intervention (ART) and suppressed HIV-1 RNA <200 copies/mL for at least 2 weeks (14 days) prior to week 24 or 48 weeks on ART (and without use of prohibited or precautionary medications based on team review of concomitant medications) were included.
Measure: Mean (95% Confidence Interval); unit: % of CD8+ T-cells
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 35
% of CD8+ T-cells | -4.01 [-6.41 to -1.61]
Statistical Analysis 1: Comparison: FTC/RPV/TDF; Estimated mean change from baseline to weeks 24-48 on ART from repeated measures (GEE) model, against the null hypothesis of zero change. Estimated mean represents on ART levels minus pre-ART levels; Test type: Other; p = 0.001, Regression, repeated measures (GEE)

2. Secondary Outcome: Plasma HIV-1 RNA Level Measured by Single Copy Assay Using Primer in Integrase (iSCA) as the Proportion of Participants Below the Limit of the Assay
Description: At a specific week, the proportion of participants with HIV-1 RNA by iSCA less than assay limit of detection (0.6 copies/mL)
Time Frame: At pre-ART and weeks 0, 4, 12, 24, 36 and 48 on ART
Population: As-treated: Only participants with results while receiving intervention (ART) and suppressed HIV-1 RNA <200 copies/mL for at least 2 weeks (14 days) prior to measured weeks on ART (and without use of prohibited or precautionary medications based on team review of concomitant medications) were included.
Measure: Number; unit: proportion of participants
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 35
proportion of participants
  Pre-ART: number analyzed (Participants) | 31
  Pre-ART | 0.19
  Week 0 on ART: number analyzed (Participants) | 31
  Week 0 on ART | 0.19
  Week 4 on ART: number analyzed (Participants) | 28
  Week 4 on ART | 0.61
  Week 12 on ART: number analyzed (Participants) | 30
  Week 12 on ART | 0.90
  Week 24 on ART: number analyzed (Participants) | 30
  Week 24 on ART | 0.93
  Week 36 on ART: number analyzed (Participants) | 26
  Week 36 on ART | 0.92
  Week 48 on ART: number analyzed (Participants) | 24
  Week 48 on ART | 0.96

3. Secondary Outcome: Change in CD4+ T-cell Count
Description: Change equals each specific week CD4+ T-cell count, respectively, minus the baseline CD4+ T-cell count (mean of the two measurements obtained prior to the start of ART)
Time Frame: From baseline (pre-ART and week 0 on ART) to weeks 12, 24, 36 and 48 on ART
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 35
cells/mm^3
  Week 12 on ART: number analyzed (Participants) | 33
  Week 12 on ART | -15 [-124 to 64]
  Week 24 on ART: number analyzed (Participants) | 33
  Week 24 on ART | -5 [-112 to 68]
  Week 36 on ART: number analyzed (Participants) | 30
  Week 36 on ART | 25 [-43 to 154]
  Week 48 on ART: number analyzed (Participants) | 29
  Week 48 on ART | 19 [-108 to 103]

4. Secondary Outcome: Change in Levels of CD8+ T-cell Activation
Description: Change equals each specific week percentage, respectively, minus the baseline percentage (mean of the two measurements obtained prior to the start of ART)
Time Frame: From baseline (pre-ART and week 0 on ART) to weeks 4, 12, 24 and 48 on ART
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: % of CD8+ T-cells
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 35
% of CD8+ T-cells
  Week 4 on ART: number analyzed (Participants) | 33
  Week 4 on ART | -0.7 [-4.7 to 4.2]
  Week 12 on ART: number analyzed (Participants) | 34
  Week 12 on ART | -1.6 [-6.2 to 4.5]
  Week 24 on ART: number analyzed (Participants) | 33
  Week 24 on ART | -2.2 [-6.1 to 0]
  Week 48 on ART: number analyzed (Participants) | 29
  Week 48 on ART | -4.7 [-7.4 to 0.3]

5. Secondary Outcome: Change in Levels of CD4+ T-cell Activation (Defined as the Percentage HLA-DR+/CD38+)
Description: as for outcome 4
Time Frame: From baseline (pre-ART and week 0 on ART) to weeks 4, 12, 24 and 48 on ART
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: % of CD4+ T-cells
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 35
% of CD4+ T-cells
  Week 4 on ART: number analyzed (Participants) | 33
  Week 4 on ART | 0.1 [-0.6 to 1.0]
  Week 12 on ART: number analyzed (Participants) | 34
  Week 12 on ART | -0.1 [-0.4 to 0.7]
  Week 24 on ART: number analyzed (Participants) | 33
  Week 24 on ART | -0.2 [-0.8 to 0.1]
  Week 48 on ART: number analyzed (Participants) | 29
  Week 48 on ART | -0.2 [-0.9 to 0.4]

6. Secondary Outcome: Change in Levels of Interleukin (IL)-6
Description: Change equals each specific week result, respectively, minus the baseline result (mean of the two log10-transformed measurements obtained prior to the start of ART)
Time Frame: From baseline (pre-ART and week 0 on ART) to weeks 4, 12, 24 and 48 on ART
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: log10(pg/mL)
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 35
log10(pg/mL)
  Week 4 on ART: number analyzed (Participants) | 33
  Week 4 on ART | 0.05 [-0.07 to 0.16]
  Week 12 on ART: number analyzed (Participants) | 33
  Week 12 on ART | 0.01 [-0.14 to 0.15]
  Week 24 on ART: number analyzed (Participants) | 32
  Week 24 on ART | 0.02 [-0.06 to 0.18]
  Week 48 on ART: number analyzed (Participants) | 27
  Week 48 on ART | 0 [-0.14 to 0.14]

7. Secondary Outcome: Change in Levels of D-dimer
Description: as for outcome 6
Time Frame: From baseline (pre-ART and week 0 on ART) to weeks 4, 24 and 48 on ART
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: log10(ng/mL)
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 35
log10(ng/mL)
  Week 4 on ART: number analyzed (Participants) | 31
  Week 4 on ART | 0.01 [-0.12 to 0.16]
  Week 24 on ART: number analyzed (Participants) | 32
  Week 24 on ART | 0.01 [-0.19 to 0.30]
  Week 48 on ART: number analyzed (Participants) | 27
  Week 48 on ART | 0.02 [-0.20 to 0.26]

8. Secondary Outcome: Change in Quality of Life (QoL) Index
Description: QoL index was obtained by averaging the five responses on the Euro-Quality of Life questionnaire (EQ-5D), where a response of 0 indicates "no problems/no discomfort", 1 indicates "some problems/moderate discomfort" and 2 indicates "unable to perform activities/extreme discomfort". Change equals each specific week index, respectively, minus the baseline index (mean of the two averages obtained prior to the start of ART)
Time Frame: From baseline (pre-ART and week 0 on ART) to weeks 4, 24 and 48 on ART
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 35
units on a scale
  Week 4 on ART: number analyzed (Participants) | 33
  Week 4 on ART | 0 [-0.1 to 0]
  Week 24 on ART: number analyzed (Participants) | 34
  Week 24 on ART | -0.1 [-0.2 to 0]
  Week 48 on ART: number analyzed (Participants) | 29
  Week 48 on ART | 0 [-0.1 to 0]

9. Secondary Outcome: Number of Subjects Who Experience Grade 3 or 4 Signs and Symptoms or Laboratory Abnormalities, Diagnoses (Any Grade), or Other Serious Adverse Events (SAEs)
Description: Grading uses the Division of AIDS (DAIDS) 2004 (clarification 2009) Severity of Adverse Events Table, where Grade 1=Mild, 2=Moderate, 3=Severe, 4=Potentially life-threatening.
Time Frame: From initiation of treatment to study completion at week 60 or 108 or premature study discontinuation
Population: All participants who initiated ART, regardless of ART status at time of event
Measure: Number; unit: participants
Arm/Group | FTC/RPV/TDF
Number analyzed (Participants) | 36
participants | 18

ADVERSE EVENTS:
Time Frame: From initiation of treatment to study completion at week 60 or 108 or premature study discontinuation
Description: The study protocol required reporting of grade>=3 signs/symptoms, grade>=3 laboratory events and all signs/symptoms and laboratory events that lead to a change in study treatment, as well as diagnoses identified by the ACTG criteria for clinical events and other diseases. See DAIDS AE Grading Table (V1.0), December 2004 (Clarification, August 2009) and EAE manual (V2.0). All participants who initiated study treatment were included.
Arm/Group | FTC/RPV/TDF
All-Cause Mortality (participants affected / at risk) | 1/36
Serious Adverse Events (participants affected / at risk) | 1/36
Other Adverse Events (participants affected / at risk) | 23/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FTC/RPV/TDF (N=36)
Bronchitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FTC/RPV/TDF (N=36)
Eye pruritus (Eye disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Proctalgia (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 2
Peripheral swelling (General disorders) | 2
Pyrexia (General disorders) | 2
Acarodermatitis (Infections and infestations) | 2
Bacterial vaginosis (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 3
Blood creatinine increased (Investigations) | 3
Blood glucose increased (Investigations) | 2
Blood phosphorus decreased (Investigations) | 5
Blood sodium decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 3
Syncope (Nervous system disorders) | 2
Vaginal discharge (Reproductive system and breast disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.